CLINICAL TRIAL: NCT00651313
Title: A Phase II, Double-Blind, Crossover Study to Assess the Efficacy and Safety of 10% (150mg) Lidocaine Vaginal Gel Administered to Women With Recurrent Dysmenorrhea
Brief Title: Efficacy and Safety Study of Lidocaine Vaginal Gel for Recurrent Dysmenorrhea (Painful Periods)
Acronym: Lidocaine 04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Juniper Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COL-1077-04
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea; Periods; Menstrual; Primary dysmenorrhea in women with recurrent dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Lidocaine 10% (150mg) vaginal gel
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Placebo vaginal gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Lidocaine vaginal gel 10% (150mg) administered once daily for 4 days
  Arms: Active
Drug: Placebo — Placebo vaginal gel administered once daily for 4 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether lidocaine vaginal gel is safe and effective for preventing or reducing the severity of dysmenorrhea (painful menstrual periods) compared to placebo (inactive gel).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of 10% (150 mg) lidocaine gel compared with placebo in reducing the severity and onset of primary dysmenorrhea in women with recurrent dysmenorrhea.

The secondary objectives of this study are the following:

* to assess the safety of 10% (150 mg) lidocaine gel compared with placebo
* to evaluate electrocardiograms (ECGs) for potentially significant QT changes at approximate peak lidocaine plasma concentration after 4 days of dosing with 10% (150 mg) lidocaine gel.

ELIGIBILITY:
Inclusion Criteria:

1. Experiences primary dysmenorrhea requiring pain medication for moderate-to-severe pain (as measured by a 4-point categorical rating scale) by the subject's own report for at least four of the previous six menstrual cycles.
2. Has a history of primary dysmenorrhea with onset within 4 years of menarche.
3. Has regular menstrual cycles (i.e. onset of menses predictable within 1 - 2 days each month) for the 3 month period preceding enrollment. If a subject has had regular cycles for the past 12 months but had a single cycle that was not regular within the 3 month period preceding enrollment, the subject may be enrolled at investigator discretion after consultation with sponsor.
4. Taking the same strength and type of hormonal contraception on a monthly cycle for at least the previous 6 months prior to screening and plans to remain on this hormonal contraception for the duration of participation in the study or is on an acceptable method of birth control including surgical sterilization (i.e. bilateral tubal ligation, partner vasectomy), double-barrier methods, and total abstinence (at the discretion of the investigator in cases where age, career, lifestyle, or sexual orientation of the patient ensures compliance).
5. Is a tampon user and/or must be willing to use tampons throughout the study dosing period.
6. Age 18 to 40 years (inclusive).
7. Has a Body Mass Index (BMI) ≤ 35 kg/m2.
8. Able to understand and willing to complete the efficacy evaluations.
9. Able to speak and understand English, and must give written informed consent for the study.

Exclusion Criteria:

1. Unable, in the opinion of the Investigator, to comply fully with any of the study requirements.
2. Experiencing pelvic pain other than that thought to be associated with primary dysmenorrhea, such as chronic pelvic pain occurring at times other than exclusively during menses and/or dyspareunia.
3. Experiencing dysmenorrhea symptoms that are effects of or thought to be effects of (at least in part) secondary causes of dysmenorrhea, such as uterine fibroids, endometriosis, and/or currently symptomatic ovarian cysts.
4. Experienced dysmenorrhea that did not require, in the opinion of the subject, the use of analgesic medication during four of the previous six menstrual episodes.
5. Has dysmenorrhea refractory to treatment with commonly used analgesic medications for the treatment of menstrual pain (e.g., ibuprofen or naproxen sodium).
6. Use of any Class I antiarrhythmic drug.
7. Currently using contraceptive injection, implant, or extended cycle OC (hormonal contraceptive cycles consisting of 28 days or more of active hormones).
8. Pregnant or breastfeeding.
9. Participated in a clinical trial in the 30 days from the time of last dosing in the prior study to the time of providing consent for this study.
10. Previously randomized into this study.
11. A history of allergic hypersensitivity or significant intolerance (including angioedema, urticaria, bronchospasm, and rhinitis) related to treatment with any medications used in this study.
12. A history of past or ongoing clinically significant disease, illness, or disorder that, in the opinion of the Investigator, makes the subject unsuitable for study participation including active vaginal, vulvar, and cervical lesions.
13. Laboratory abnormalities that, in the opinion of the Investigator, could contraindicate study participation such as liver function tests > 1.5 times the upper limit of normal (At the Investigator's discretion, laboratory tests may be repeated once for verification.)
14. A history of, within the past 4 years, or ongoing significant psychiatric illness that, in the opinion of the Investigator, makes the subject unsuitable for study participation.
15. A history of chronic analgesic or tranquilizer use or drug abuse including alcohol within the 6 months before providing consent for this study.
16. Regular use of any concomitant medications that might confound efficacy and/or safety assessments, in the opinion of the Investigator, including, but not limited to, the following: psychotropic drugs, antidepressants, sedative-hypnotics, sedating antihistamines, or tranquilizers for 24 hours or five half-lives prior to providing informed consent until 24 hours after the final treatment cycle. Selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), and St. John's Wort are permitted for indications other than pain if the subject has been on a stable dose for at least 2 weeks before providing consent for this study and agrees to remain on a stable dose throughout the course of the study.
17. Unwilling to use only those medications that are allowed in the study for the treatment of their dysmenorrhea, i.e., study drug and rescue medication.
18. Any ongoing vaginal infection requiring intravaginal treatment.
19. A history of toxic shock syndrome (TSS).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George W Creasy, MD, Study Director — Juniper Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - SCIREX Research Center, Memphis, Tennessee
  - SCIREX Research Center, Austin, Texas
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinics and private practice offices; 8/31/07-6/13/08. Maximum patient participation was approx 4 months, including 45 day screening period, a treatment period of approx 8 weeks duration (during which subjects received study drug on a total of 8 days), and a post treatment visit occurring 2 - 3 weeks after Treatment Cycle 2,Visit 5.
Pre-assignment Details: Crossover study; Subjects who met study entry criteria after completing screening procedures at Screening Visit returned to study center at least 7 days prior to their expected onset of menses to complete Randomization/Treatment procedures. Abnormal lab values, ECGs or use of prohibited medications were among reasons subjects were excluded.
Period: Overall Study
Arm/Group | Active | Placebo
Started | 41 | 43
Completed | 35 | 37
Not Completed | 6 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adminstrative Discontinuation | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 43 | 84
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.5 (7.20) | 27.7 (6.69) | 27.1 (6.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 84
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Variable Will be the Time-weighted Average Pain Intensity Over 4 Treatment Days Using the 4 Point Categorical Scale.
Time Frame: Two 4-day dosing regimens for two consecutive monthy menstrual cycles
Population: Time-weighted average pain intensity over the 4 treatment days using the 4 point categorical scale - none (0), mild (1), moderate (2), and severe (3); primary efficacy variable. ITT Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lidocaine 10%; Placebo Gel: Crossover Study Sequence 1 = 10% Lidocaine Gel to Placebo Gel Sequence 2 = Placebo Gel to 10% Lidocaine Gel
Arm/Group | Lidocaine 10% | Placebo Gel
Number analyzed (Participants) | 70 | 70
units on a scale | 0.91 (0.635) | 0.92 (0.552)

2. Primary Outcome: Treatment-emgergent Adverse Events
Time Frame: approximately two months, based on onset of menses
Reporting Status: Not Posted

3. Secondary Outcome: Evaluate Electrocardiograms (ECGs) for Potentially Significant QT Changes at Approximate Peak Lidocaine Plasma Concentration After 4 Days of Dosing
Time Frame: 7 hours following fourth dose in 2 consecutive menstrual cycles
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 6/77 | 7/77
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=77) | Placebo (N=77)
Headache (Nervous system disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days